CLINICAL TRIAL: NCT04881422
Title: Sport, Rehabilitation and Nutrition in Multiple Sclerosis: An Innovative Multidisciplinary High Impact Intervention for the Lifestyle Change
Brief Title: Sport, Rehabilitation and Nutrition in Multiple Sclerosis: The LINUS Project
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07_23/05/2018
Record Dates: First submitted 2021-04-28; First posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Multiple Sclerosis
Keywords: lifestyle; multiple sclerosis; nutrition; rehabilitation; motivation; adherence
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): A group of pwMS participate in a multidimensional integrate high-motivating rehabilitation program for the change of lifestyle and bad habits.
  Interventions: Behavioral: B-HIPE (Brief High Impact Preparatory Experience)

INTERVENTIONS:
Behavioral: B-HIPE (Brief High Impact Preparatory Experience) — The intervention consists in a one-week intensive rehabilitation in which participants underwent to a multidimensional rehabilitation composed by physical rehabilitation, mental wellbeing, a proper diet and engaging physical activity (a sail course). Digital motivating reinforcements are proposed to the participants with the aim to maintain the correct lifestyle learned in the B-HIPE program.

SUMMARY:
Only a limited percentage of persons with MS (pwMS) participate to multidisciplinary rehabilitation because of poor support, knowledge and motivation. The investigators reasoned that pwMS should be more effectively prepared to increase their adherence. This study propose the implementation of an innovative collaborative approach, called "brief high-impact preparatory experience" (b-HIPE), inspired by an overarching model based on the interplay between competence, motivation and opportunity to increase in a short time awareness and motivation of pwMS.

The aim of the study is the evaluation of its feasibility. For this pilot study the investigator chose a single-group design with repeated measurements at baseline and post intervention.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 70 years
* EDSS ranging from 1 to 7.5.
* pwMS with who are on a western diet
* stabilized medical therapy and clinical conditions
* pwMS with a motor control of upper limbs sufficient to maneuver a tiller

Exclusion Criteria:

* Heavy smoking, alcohol and drugs abuse
* severe cognitive impairment
* dysphagia and/or comorbidities requiring protected environments and specific medical assistance
* blindness and severe visual disturbances (included severe nystagmus)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-07-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
FS-36 Health Related Quality of Life (HRQoL) | Change between the baseline - T0 (before the intervention) and 1 month after the end of the intervention (T1)
  Questionnaire to Measure Health-Related Quality of Life
The Fatigue Severity Scale (FSS) | Change between the baseline - T0 (before the intervention) and 1 month after the end of the intervention (T1)
  Questionnaire to Measure the fatigue
Food frequency questionnaire (FFQ) | Change between the baseline - T0 (before the intervention) and 1 month after the end of the intervention (T1)
  Questionnaire to evaluate usual frequency of foods and beverages

SECONDARY OUTCOMES:
MSIS29- Multiple Sclerosis Impact Scale | Change between the baseline - T0 (before the intervention) and 1 month after the end of the intervention (T1)
  A scale for the evaluation of the impact of MS on day-to-day life
MOS Sleep Scale (MOSS) | Change between the baseline - T0 (before the intervention) and 1 month after the end of the intervention (T1)
  A scale for the evaluation of the quality and the quantity of sleep
Restless Legs Scale (RLS) | Change between the baseline - T0 (before the intervention) and 1 month after the end of the intervention (T1)
  A scale for the evaluation of the restless legs syndrome
Six minute walking test (6MWT) | Change between the baseline - T0 (before the intervention) and 1 month after the end of the intervention (T1)
  An exercise test used to assess aerobic capacity and endurance
Hospital Anxiety and Depression Scale (HADS) | Change between the baseline - T0 (before the intervention) and 1 month after the end of the intervention (T1)
  A self-assessment scale for detecting states of depression and anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi, Milan, Italy